CLINICAL TRIAL: NCT03333798
Title: A Cognitive-Behavioral Intervention With Community Worker Support for Survivors of Intimate Partner Violence in Cali and Tuluá, Colombia.
Brief Title: Psychosocial Intervention With Community Worker Support for Survivors of Intimate Partner Violence
Acronym: IPCCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Universidad Unidad Central del Valle (UCEVA) (Unknown); Red de Salud de Ladera E.S.E (Unknown); Hospital Rubén Cruz Vélez E.S.E (Unknown); Heartland Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Code No.110674456022
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Intimate Partner Violence; Depression; Anxiety; Post-traumatic Stress Disorder; Activities of Daily Living; Self Esteem
Keywords: Intimate Partner Violence; Domestic Violence; Mental Health; Cognitive- Behavioral Therapy; Community Lay Workers
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-Behavioral Intervention (Experimental): Cognitive-Behavioral Intervention with community worker support.
  Interventions: Behavioral: Cognitive-Behavioral Intervention
- Standard psychosocial care (Active Comparator): Standard psychosocial care delivered by health services.
  Interventions: Behavioral: Standard psychosocial care

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Intervention — A Cognitive-Behavioral intervention will be delivered by psychologists with LPCWs support. LPCWs who will be under the supervision and guidance of psychologists.
  Volunteers will receive 11 weekly sessions of which six will be provided by psychologists and five by LPCWs.
  The Cognitive-Behavioral component will be delivered through a set modules that will cover the following components:
  * The Cognitive-Behavioral model
  * Tackling traumatic events
  * Cognitive reprocessing
  * Relaxation techniques
  * Prevention of revictimization
  * Behavioral reactivation for the start of a new life The intervention will be given within the health system and volunteers will be seen if necessary by an interdisciplinary team including social workers, general physicians and psychiatrists.
  Arms: Cognitive-Behavioral Intervention
Behavioral: Standard psychosocial care — The active control group will receive standard psychosocial care for intimate partner violence, provided by the participating health centers. Standard care is delivered by psychologists, social workers, general physicians and psychiatrists. Additionally, patients receive extramural support which includes telephone calls or domiciliary visits from a variety of health professionals (doctors, nurses, social workers and nursing assistants).
  Psychology consultations typically occur every four weeks in each health center. Psychologists use a variety of approaches according to their personal preferences, including humanist, psychoanalytic, psychodynamic and cognitive-behavioral approaches. At the end of the intervention psychologists will be asked which approach or approaches they used.
  Arms: Standard psychosocial care

SUMMARY:
Female survivors of domestic violence (DV) may exhibit various mental health problems. A variety of psychotherapies are available to improve their mental health, however there is uncertainty on which is the best. In Colombian, national guidelines do not mention which therapy should be used and in practice, psychologists use their preferred approaches. Due to the shortage of psychotherapy appointments, patients wait a long time to initiate treatment and for each subsequent appointment. Furthermore, patients with mental health problems often fail to attend their appointments and often drop-out of their psychotherapy. This study will offer an alternative intervention that is hypothesized to be superior to normal patient care in Colombia. It will be conducted in Cali and Tuluá, which have high levels of DV, internally displaced conflict victims and large socioeconomic inequalities. Psychologists and trained Lay Psychosocial Community Workers (LPCWs) will work together to provide a cognitive-behavioral intervention (CBI) for female survivors of DV, which is a therapy that aims to change the way people think and behave. Each woman will be offered 11 weekly sessions which will be shared between a psychologist and a LPCW. The LPCW will assign tasks to the patients which have been set by the psychologist and will assist participants to attend their appointments. The study´s hypothesis is: 1) A psychologist led CBI with LPCW support is superior to standard psychotherapy care in Colombian health services to improve mental health symptoms of female survivors of DV.

Patients will be recruited from health services and will be randomly assigned to either the standard psychotherapy or the CBI with LPCW support (intervention group). In the standard psychotherapy group, patients will receive psychotherapy approximately every four weeks, depending on demand, and will have as many sessions as they require. In the intervention group, patients will be offered eleven weekly CBI sessions. Mental health questionnaires will be used to measure the study participants' mental health symptoms, their functionality, experience of DV and other forms of violence. In the intervention group, these questionnaires will be applied before initiating psychotherapy, two weeks and six months after completing their psychotherapy. Patients in the control group will have questionnaires applied before commencing psychotherapy and fourteen weeks and twenty-two weeks after starting.

DETAILED DESCRIPTION:
Intimate partner violence (IPV) is a complex problem because it is associated with factors at a variety of levels which include the individual, conjugal, societal, cultural, and institutional, which can all also act as barriers to accessing mental health services. Survivors of IPV are vulnerable to an array of mental health illnesses which include post-traumatic stress disorder (PTSD), depression, anxiety, emotional dependency and low self-esteem. A variety of psychotherapies are available to improve mental illnesses, however there is uncertainty on which is the superior approach. In Colombia there are no national guidelines outlining which therapy should be used, rather, psychologists use their preferred approach or approaches which may include humanistic or psychoanalytical methods. Furthermore, patients with mental health problems face a large waiting list for initial and follow-up psychotherapy appointments, often fail to attend and do not complete their treatment. This study will be conducted in two cities, Cali and Tuluá, in the state Valle del Cauca that have high levels of IPV, internally displaced conflict victims and large socioeconomic inequalities.

The study´s hypothesis is that a psychologist led cognitive-behavioral intervention with Lay Psychosocial Community Worker (LPCW) support is superior to treatment as usual to reduce mental illness symptoms. The study's objective is to improve mental illness symptoms of female survivors of IPV through the program IPCCOS, a Cognitive-Behavioral Intervention with Community Worker Support for Survivors of Intimate Partner Violence (IPCCOS is the abbreviation for its name in Spanish: Intervención Psicoterapéutico Cognitivo-Conductual con Apoyo Comunitario para Sobrevivientes de Violencia de Pareja). IPCCOS was developed by the CISALVA Institute at the Universidad del Valle (Cali), the Universidad Central del Valle del Cauca UCEVA (Tuluá), with assistance from Heartland Alliance International (HAI) to provide and test an alternative intervention for female survivors of IPV. Each patient will be offered 11 weekly psychotherapy sessions which will be divided between a psychologist and a LPCW. The LPCWs in the study will come from community women groups who are already working in women´s rights and have exposure to violence against women and the relevant medico-legal systems. They will receive up to a week of intensive training from study psychologists and a psychologist from HAI who is trained in cognitive-behavioral therapy (CBT) and has experience training and supervising LPCWs in other mental health studies in Colombia. Approximately six weeks after initiating the intervention, LPCWs will receive a further day of training. LPCWs will assign tasks to patients which have been set by the psychologist and will assist them to overcome any barriers to attend their appointments. They will be closely supervised by the psychologist once per week to discuss their patients.

A randomized control trial study design will be used to compare and evaluate the two groups. Patients will be recruited from health services if they are found to have experimented IPV in the last year and will be randomly assigned by block randomization to either treatment as usual or the IPCCOS (intervention group). Patients will be invited to participate in the study from three sources:

* General physician outpatient appointments.
* Hospital data bases. Hospital records will be searched to detect patients that have experienced IPV and that have not commenced psychotherapy. This will be performed retrospectively to search for patients that were given this diagnosis of IPV between January 2017 and September 2017. They will be contacted via phone, given a brief description of the study and if they are interested in participating, they will be invited to meet a health professional who will give a more detailed description of the study and take informed consent.
* Patients that are detected to have experienced IPV in the Emergency Department will be told about the study. They will only be asked to decide on their participation one week after they have been discharged.

In the treatment as usual group, patients normally receive psychotherapy every four weeks, depending on demand. There is no pre-established number of sessions as this depends on the clinical condition and the patient´s adherence.

In the intervention group, patients will be offered eleven weekly cognitive-behavioral sessions that will be delivered by psychologists and LPCWs. In addition, they will receive phone calls from LPCWs to remind them of their appointments.

The sessions will be divided between psychologists and LPCWs in the following scheme:

1. Psychologist
2. Psychologist
3. Psychologist
4. LPCW
5. LPCW
6. Psychologist
7. LPCW
8. LPCW
9. Psychologist
10. LPCW
11. Psychologist

LPCWs will meet with psychologists on a weekly basis to discuss their patients and any safety concerns.

Patients who exhibit severe mental illness symptoms during the intervention such as suicidal ideation, schizophrenia or bipolar disorder will be referred to the project psychiatrist for specialist care.

An array of instruments will be applied during the study to measure mental illness symptoms, functionality, IPV experience and other forms of violence. These measures will be taken immediately before starting psychotherapy and two weeks and six months after completing the intervention in the intervention group. Patients in the control group will have instruments applied before commencing psychotherapy and fourteen weeks and twenty-two weeks after starting.

Sample size:

A sample size was calculated according to the following formula (comparison of means from the intervention and control groups):

n = 2 (Zα + Zβ)² * S² (x1 - x2) ²

The sample size was calculated using values from a previous cognitive-behavioral intervention for armed-conflict victims of Buenaventura and Quibdó, Colombia (https://clinicaltrials.gov/ct2/show/NCT01856673). An Alfa error of 5%, power of 80%, and standard deviation of 30 was used. The sample size of each arm necessary to obtain a significant difference in means of symptoms between the control and intervention group is:

n = 2 (1.96 + 0.842)² * 30² / (20) ²

n = 35

According to this calculation a minimum of 35 volunteers must be recruited into each arm per city (Cali and Tuluá), which means that overall 70 volunteers will be recruited into the intervention group and 70 volunteers into the control group giving a total of 140 volunteers in the study.

Information will be collected using digital tablets and transferred to a database designed for the study. Confidentiality will be ensured by not including identifying variables.

An exploratory analysis to identify extreme values or missing data will be performed and medical records will be revised to verify some of the information. A sample of the instruments applied in the study will be audited.

Multiple imputation techniques will be used for all missing data including those resulting from lost to follow up. Additionally, a sensitivity analysis based on probability weighting will be used as a covariate in the final analysis for all missing data.

The anticipated results are a reduction in anxiety, depression, PTSD, low self-esteem and emotional dependency symptoms, which will be greater in patients in the intervention group compared those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Female survivors of IPV
* Inhabitants of Cali or Tuluá, Valle del Cauca
* 18 years old or older

Exclusion Criteria:

* Severe mental illness that requires specialized treatment (determined by a psychiatrist or psychiatry resident)
* Terminally ill
* Decompensated chronic diseases
* Hypothyroidism (not controlled by medication)
* Neurosyphilis
* Under psychiatric medication
* Sexual abuse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Score Difference in Symptoms of Anxiety | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Anxiety symptoms will be assess using the Hopkins Symptom Checklist (HSCL-25)
Score Difference in Symptoms of Depression | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Depression symptoms will be assess using the Hopkins Symptom Checklist (HSCL-25)
Score Difference in Symptoms of Post-Traumatic Stress Disorders | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Symptoms of trauma (PTSS) will be assess using the Harvard Trauma Questionnaire (HTQ).

SECONDARY OUTCOMES:
Score Difference in Disability | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Disability will be assess using the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0).
Score Difference in Self-Esteem. | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Self-esteem will be assess using the Rosenberg's Self-Esteem Scale. Each question has response that gives a score between 1-4. A mean score of responses will be calculated to give the final score.
Score Difference in Emotional Dependence Scales. | Measurement at baseline before the intervention, and within the fifteen (15) days after finishing the intervention. In the control group, 12 weeks after the baseline assessment.
  Emotional dependency will be asses using the Emotional Dependence Scale (Cuestionario de Dependencia Emocional). Each question has response that gives a score between 1-6. A mean score of responses will be calculated to give the final score.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Fandiño, MD, PhD, Principal Investigator — Universidad del Valle

IPD SHARING:
Plan to Share IPD: No
Not planned.

REFERENCES:
- [Background] Murray LK, Dorsey S, Bolton P, Jordans MJ, Rahman A, Bass J, Verdeli H. Building capacity in mental health interventions in low resource countries: an apprenticeship model for training local providers. Int J Ment Health Syst. 2011 Nov 18;5(1):30. doi: 10.1186/1752-4458-5-30. PMID 22099582
- [Background] Johnson DM, Zlotnick C, Perez S. Cognitive behavioral treatment of PTSD in residents of battered women's shelters: results of a randomized clinical trial. J Consult Clin Psychol. 2011 Aug;79(4):542-551. doi: 10.1037/a0023822. PMID 21787052
- See also: Evaluation of Two Community-based Mental Health Interventions for Violence-Displaced Afro-Descendants in Colombia. (ACOPLE) — https://clinicaltrials.gov/ct2/show/NCT01856673